CLINICAL TRIAL: NCT02280109
Title: Comparison of the Pharmacokinetics and Pharmacodynamics of Single Dose Tenofovir Vaginal Gel and Film Formulation
Brief Title: Comparison of Tenofovir Vaginal Gel and Film Formulations
Acronym: FAME-05
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Craig Hendrix, Professor of Medicine, Pharmacology and Molecular Sciences, Division of Clinical Pharmacology Johns Hopkins University School of Medicine, CONRAD
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DAIDS-ES #12015; U19AI082639 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-31 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Healthy; HIV
Keywords: Tenofovir; Healthy Volunteers; HIV; pharmacokinetics of tenofovir gel and film
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir Gel (Active Comparator): Women will receive a single dose of tenofovir gel (1%;equivalent to 40 mg in 4ml's of gel) to determine the pharmacokinetics of tenofovir in the blood, cervical tissue, and cervicovaginal fluid.
  Interventions: Drug: Tenofovir Gel
- Tenofovir Film (Active Comparator): Women will receive a single dose of tenofovir film (1.3%;40 mg) to determine the pharmacokinetics of tenofovir in the blood, cervical tissue, and cervicovaginal fluid.
  Interventions: Drug: Tenofovir Film

INTERVENTIONS:
Drug: Tenofovir Gel — single dose of 1% tenofovir gel (equivalent to 40 mg in 4ml's of gel)
  Other Names: Tenofovir disoproxil
  Arms: Tenofovir Gel
Drug: Tenofovir Film — single dose of 1.3% tenofovir film (equivalent to 40 mg)
  Other Names: Tenofovir disoproxil
  Arms: Tenofovir Film

SUMMARY:
This is an open label comparative study of tenofovir gel and film in 10 healthy sexually active women without active female genital tract disorders. The women will receive a single dose of each formulation - tenofovir gel (1%;equivalent to 40 mg in 4ml's of gel) and tenofovir film (1.3%;40 mg) - in a crossover study design to determine the pharmacokinetics of tenofovir in the blood, cervical tissue, and cervicovaginal fluid (primary objective).

DETAILED DESCRIPTION:
This is an open label comparative study of tenofovir gel and film in 10 healthy sexually active women without active female genital tract disorders. The women will receive a single dose of each formulation - tenofovir gel (1%;equivalent to 40 mg in 4ml's of gel) and tenofovir film (1.3%;40 mg) - in a crossover study design to determine the pharmacokinetics of tenofovir in the blood, cervical tissue, and cervicovaginal fluid (primary objective). Further, pharmacodynamics will be assessed using cervical tissue in an ex vivo HIV biopsy challenge, and safety will be determined by assessment of adverse events following a single dose of each formulation (secondary objective). The primary endpoint will be to determine concentrations of tenofovir (TFV) and its metabolite, tenofovir diphosphate (TFV-DP), in plasma, tissue homogenates, and cervicovaginal fluid. Secondary endpoints will be determined by assessing concentrations of HIV p24 protein from explant aliquot samples up to 21 days post-infection ex vivo, and by determination of Grade 2 or higher adverse events deemed related to study product.

Research participants will receive the first tenofovir dose formulation prior to the following sampling:

* Blood PK plasma collection will be obtained at pre-dose, 0.5, 1, 2, 4, 5, 8 and 12 hours (Day 0), 24 hours (Day 1); 48 hours (Day 2); 72 hours (Day 3); and 168 hours (Day 7) following tenofovir formulation dosing.
* Cervicovaginal fluid sampling, rectal fluid sampling, and cervicovaginal biopsy will be performed (in the sequence listed) 5 and 72 hours after dosing in all subjects. Cervicovaginal fluid and rectal fluid sampling will also be obtained at 168 hours.

Subjects will be counseled to abstain from sexual intercourse and all other insertive vaginal practices for 10 days following each administered dose (or 7 days after the last cervicovaginal sampling at 72 hours). Following a safety evaluation visit, the research participant will return to the research unit and receive a second tenofovir dose formulation followed by the same schedule of sample collection and a final safety visit. PK parameters of TFV and TFV-DP will be estimated and compared between the gel and film formulations. PK parameters will include peak concentration (Cmax), area under the concentration-time curve (AUC), time to peak concentration (Tmax), elimination half-life (t1/2). Tenofovir gel and film ex vivo pharmacodynamics will also be assessed and analyzed for correspondence to pharmacokinetics.

Visit 1 Visits 2-6 Visit 7 Visits 8-12 Visit 13

- 28 Days Day 0-7 Day 14 Day 28-35 Day 42

These studies will be carried out at The Johns Hopkins Hospital under the direction of Craig Hendrix, MD, as the Project PI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years of age (inclusive) with a history of receptive vaginal intercourse.
2. HIV negative within 28 days of enrollment
3. Understand and agree to local STI reporting requirements.
4. Able and willing to provide written informed consent to take part in the study.
5. Able and willing to provide adequate information for locator purposes.
6. Availability to return for all study visits, barring unforeseen circumstances.
7. Availability to return for the second formulation dosing at the same time in the subject's menstrual cycle as when the first formulation was administered, at least 10 days before menses.
8. Willing to abstain from vaginal intercourse and insertion of anything (e.g., drug, vaginal douche, personal lubricant or sex toy) in vagina for 72 hours before each study product exposure, and 10 days following study product dosing, comprising a total of 26 days of abstinence, no insertion of vaginal products/objects while participating in the study.
9. Willingness to have partner(s) use condoms (must not contain Nonoxynol-9) for the duration of the study.
10. Agree not to participate in other research studies involving drugs and/or medical devices.
11. Negative qualitative urine pregnancy test.
12. Using an effective method of contraception at enrollment.
13. Willingness to remain in the research unit for up to 12 hours on each of two dosing days.

Exclusion Criteria:

1. Current sexual partner known by participant to be HIV seropositive.
2. Individuals who, by history, engage in condom-less intercourse with HIV-infected partners, or partners that have unknown HIV serostatus, or women who exchange sex for money, shelter, or gifts.
3. Active chlamydia, gonorrhea, syphilis, trichomonas, cervicitis or PID within 8 weeks prior to enrollment.
4. Individuals with active hepatitis B infection.
5. Known history of genital HSV (diagnosed by either clinical or laboratory test).
6. Symptomatic vaginal candidiasis or bacterial vaginosis.
7. Undiagnosed irregular uterine bleeding
8. Pathology of the female genital tract,
9. Individuals who are status post hysterectomy.
10. History of any cervicovaginal procedure (i.e. colposcopy with cervical biopsy) within the past 2 months.
11. History of cone biopsy or extensive loop electrosurgical excision procedure (LEEP), which in the judgment of the investigator may affect permeability assessment.
12. Any known primary or secondary uro-genital malformations, which in the assessment of the investigator may interfere with the intended urine collection for PK studies.
13. Use of vaginally administered medications within 4 week of enrollment
14. Any active urinary tract infection
15. By history, subjects with irregular menstrual cycles.
16. At screening:

    * ALT or AST greater than 1.5 X the site laboratory ULN
    * Hemoglobin less than 10.0 g/dL
    * Platelet count less than 100,000/mm3
    * Other safety tests outside of the normal range
    * Findings that are clinically significant in the opinion of the investigator
17. Estimated creatinine clearance < 60 ml/min based on established nomograms
18. Recent history (past 6 months) of injection drug use or alcohol use that may interfere with the study.
19. Unwillingness to refrain from aspirin and NSAIDs product use for one week prior to and one week post study procedures.
20. Use of warfarin or heparin.
21. Use of systemic immunomodulatory medications within 4 weeks of enrollment.
22. Use of product containing nonoxynol-9 within 4 weeks of enrollment.
23. Use of any investigational products within 4 weeks of enrollment.
24. Any other medical conditions deemed not safe for participation by the investigator.
25. Any individual that is pregnant or is actively breast feeding.
26. Post-menopausal defined as 12 months of amenorrhea.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma tenofovir concentration-time curve (AUC0-72) for each product (film and gel) 0 thru 72 hours after dosing | 72 hours
  Concentration-time plot of plasma tenofovir
PBMC tenofovir diphosphate concentration-time curve (AUC0-72) for each product (film and gel) 0 thru 72 hours after dosing | 72 hours
  Concentration-time plot of PBMC tenofovir diphosphate thru 72 hours after dosing
Cervical tissue tenofovir maximum concentration (Cmax) at 5 hours | 5 hours
Cervical tissue tenofovir maximum concentration (Cmax) at 72 hours | 72 hours
Cervical tissue tenofovir diphosphate maximum concentration (Cmax) at 5 hours | 5 hours
Cervical tissue tenofovir diphosphate maximum concentration (Cmax) at 72 hours | 72 hours
Cervicovaginal fluid tenofovir maximum concentration (Cmax) at 5 hours | 5 hours
Cervicovaginal fluid tenofovir maximum concentration (Cmax) at 72 hours | 72 hours
Rectal fluid tenofovir maximum concentration (Cmax) at 5 hours | 5 hours
Rectal fluid tenofovir maximum concentration (Cmax) at 72 hours | 72 hours
All adverse clinical and laboratory events | one year
  Categorize adverse events by treatment formulation to compare the safety of single dose tenofovir gel and film formulations

SECONDARY OUTCOMES:
Cumulative HIV p24 protein concentration from 0 to 15 days post ex-vivo infection of explant cervical tissue collected at 5 hours after dosing with tenofovir gel or film | 15 days
Cumulative HIV p24 protein concentration from 0 to 15 days post ex-vivo infection of explant cervical tissue collected at 72 hours after dosing with tenofovir gel or film | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Craig W Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine Division of Clinical Pharmacology, Baltimore, Maryland, United States